CLINICAL TRIAL: NCT00656630
Title: Medication Development in Protracted Abstinence in Alcoholism: Acamprosate Versus Naltrexone
Brief Title: Medication Development in Alcoholism: Acamprosate Versus Naltrexone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AA012602; R01AA012602 (NIH)
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate; Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Acamprosate
  Interventions: Drug: Acamprosate
- 2 (Active Comparator): Naltrexone
  Interventions: Drug: Naltrexone
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acamprosate — Two 333mg capsules, 3 times daily (Total dose, 1998 mg daily), 1 week duration
  Other Names: Campral
  Arms: 1
Drug: Naltrexone — 50mg capsule, Once daily, 1 week duration
  Other Names: ReVia
  Arms: 2
Drug: Placebo — Matched placebo capsule, 1 week duration
  Other Names: Sugar pill
  Arms: 3

SUMMARY:
The purpose of this study is to develop and validate a human laboratory model for prediction of medication efficacy in clinical trials for relapse prevention in alcohol dependence.

DETAILED DESCRIPTION:
This is a double-blind, 3-cell, outpatient human laboratory study to determine the degree to which acamprosate and naltrexone will suppress subjective and physiological responsivity to alcohol cues relative to placebo in early abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 and ≤ 55 years of age
* Meets Diagnostic and Statistical Manual-Fourth Edition (DSM-IV) criteria for current alcohol dependence
* Does not desire treatment
* Alcohol free, as verified by breath alcohol concentration, with a Clinical Institute Withdrawal Assessment (CIWA) ≤ 8, at the time of testing, with no evidence of drinking for at least 3 days but no more than 7 days prior to the cue reactivity session
* Able to complete and understand questionnaires and study procedures in English
* Verbal I.Q. estimate ≥ 85
* Signed informed consent

Exclusion Criteria:

* Currently meets DSM-IV criteria for dependence on substances other than alcohol or nicotine
* Significant medical disorders that will increase potential risk or interfere with study participation
* Sexually active women with childbearing potential who are pregnant, nursing, or refuse to use a reliable method of birth control
* Meets DSM-IV criteria for a major Axis I disorder, including depression or anxiety disorders
* Treatment within the month prior to screening with investigational medications or those which may influence drinking outcome, e.g., disulfiram (Antabuse), naltrexone (ReVia), acamprosate (Campral), antidepressants or other psychotropic agents
* Chronic treatment with any narcotic-containing medications during the previous month or evidence of current opiate use
* Liver function tests more than three times normal or elevated bilirubin
* No fixed domicile and/or no availability by telephone or beeper
* Current involvement in or plans for treatment prior to study completion
* Patients who have a history of adverse drug reactions to the study drugs or their ingredients
* Failure to take double-blind medication as prescribed
* Inability to understand or comply with the provisions of the protocol or consent form

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study participation at the Laboratory of Clinical Psychopharmacology at The Scripps Research Institute in La Jolla, California from 04/17/2008-12/10/2009. Sixty eight subjects were enrolled, and sixty two subjects completed the study.
Groups:
- Campral (Acamprosate): Acamprosate
  Acamprosate: Total dose, 1998 mg daily, 1 week duration
- ReVia (Naltrexone): Naltrexone
  Naltrexone: 50mg capsule, Once daily, 1 week duration
- Sugar Pill (Placebo): Placebo: Double-dummy placebo capsules, 1 week duration
Period: Overall Study
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo)
Started | 22 | 27 | 19
Completed | 20 | 25 | 17
Not Completed | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo) | Total
Number analyzed (Participants) | 22 | 27 | 19 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.73 (10.10) | 36.37 (12.45) | 42.84 (10.37) | 37.97 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 6 | 22
  Male | 12 | 21 | 13 | 46
Region of Enrollment [Number; unit: participants]
  United States | 22 | 27 | 19 | 68

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale of Craving to Drink at 1 Week Following Administration of Acamprosate or Naltrexone or Placebo During the Double-Blind Period
Description: The four Visual Analog Scale questions assess domains of alcohol craving: the intention to drink, loss of control, relief craving, and urge intensity. The scale ranges from 0-20 where a zero indicates no craving and 20 indicates severe craving; thus, a higher score indicates a worse outcome. Total is a summation of the four subscales (i.e. Strength, Intent, Impulse, Relief) and ranges in value from 0-80 with higher scores indicative of a worse outcome.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo)
Number analyzed (Participants) | 20 | 25 | 17
units on a scale
  Strength | 2.12 (3.10) | 3.40 (3.87) | 5.86 (4.79)
  Intent | 1.65 (1.56) | 2.99 (3.67) | 4.22 (4.34)
  Impulse | 1.17 (1.94) | 1.69 (2.78) | 4.31 (4.82)
  Relief | 0.07 (1.67) | 2.01 (3.56) | 3.57 (4.14)
  Total | 5.00 (6.24) | 10.09 (12.12) | 17.96 (15.83)

2. Secondary Outcome: Change From Baseline in Standard Drinks Per Week at 1 Week
Description: Standard drinks are equivalent to 14 grams of pure alcohol and number of drinks are assessed with Timeline Follow-Back (TLFB) methods. Change = (Week 1 - Baseline). More negative values indicate less use of alcohol.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: drinks/week
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo)
Number analyzed (Participants) | 20 | 25 | 17
drinks/week
  Drinks/week Baseline | 44.90 (61.89) | 47.02 (24.08) | 48.87 (58.53)
  Drinks/week Week 1 | 24.37 (22.81) | 25.79 (14.32) | 21.51 (18.88)
  Drinks/week Change | -20.53 (60.68) | -21.23 (23.93) | -27.35 (44.84)

3. Secondary Outcome: Change From Baseline in Mood on the Beck Depression Inventory (BDI-II) at Week 1
Description: The BDI-II is a self-rating of severity of depressive symptoms. BDI-II Total scores range from 0-63; a lower score indicates less severe depressive systems and thus is a better outcome. Change = (Week 1 score - Baseline score). The Total score is a sum of the 21 items on the BDI-II instrument, with each item rated from 0-3.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo)
Number analyzed (Participants) | 20 | 25 | 17
units on a scale
  BDI-II Total Baseline | 4.40 (5.14) | 4.04 (4.33) | 3.53 (4.74)
  BDI-II Total Week 1 | 4.75 (4.81) | 3.84 (4.02) | 4.94 (5.70)
  BDI-II Total Change | 0.35 (4.16) | -0.20 (2.84) | 1.41 (4.30)

4. Secondary Outcome: Change From Baseline in Sleep Quality on the Pittsburgh Sleep Quality Index (PSQI) Total Score at Week 1
Description: The PSQI is an instrument to assess subjective sleep quality and disturbance. The Total score ranges from 0 to 21 where a lower score is better sleep quality. Change = (Week 1 score - Baseline score). Seven subscales (range 0-3) are summed to compute the Total score.
Time Frame: 1 week
Population: Seven participants who completed the double blind portion of the trial were unable to be analyzed for change in PSQI Total score due to incomplete PSQI questionnaire at baseline and/or Week 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo)
Number analyzed (Participants) | 16 | 23 | 16
units on a scale
  PSQI Total Baseline | 4.50 (3.14) | 4.74 (3.62) | 4.25 (2.82)
  PSQI Total Week 1 | 4.69 (3.88) | 4.57 (3.55) | 4.38 (3.67)
  PSQI Total Change | 0.19 (3.78) | -0.17 (2.08) | 0.13 (2.68)

5. Secondary Outcome: Change From Screening in Craving on the Alcohol Craving Questionnaire-Short Form (ACQ-SF) Total Score at Week 1
Description: The ACQ-SF is an assessment of current drinking urges, difficulty resisting urge and anticipation of positive outcome or relief from negative state by drinking. The Total score ranges from 0 to 7 where a lower score is a better outcome. Change = (Week 1 score - Screening score). The scale is comprised of twelve items (range 0-7) that are averaged to compute the Total score.
Time Frame: 2 weeks
Population: One participant in the naltrexone arm who completed the double blind portion of the trial was unable to be analyzed for change in ACQ-SF Total score due to incomplete ACQ-SF questionnaire at Week 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Campral (Acamprosate) | ReVia (Naltrexone) | Sugar Pill (Placebo)
Number analyzed (Participants) | 20 | 24 | 17
units on a scale
  ACQ-SF Total Screening | 3.80 (1.38) | 3.81 (1.55) | 3.99 (1.34)
  ACQ-SF Total Week 1 | 3.36 (1.28) | 3.69 (1.26) | 3.51 (0.98)
  ACQ-SF Total Change | -0.44 (1.02) | -0.12 (1.56) | -0.48 (1.12)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all four study visits, an average duration of 4 weeks.
Description: Adverse events, both serious and other, were documented at all four study visits by the Medical Assistant on the adverse event case report form.
Groups:
- Acamprosate: Acamprosate
  Acamprosate: Total dose, 1998 mg daily, 1 week duration
- Naltrexone: Naltrexone
  Naltrexone: 50mg capsule, Once daily, 1 week duration
- Placebo: Placebo: Double-dummy placebo capsules, 1 week duration
Arm/Group | Acamprosate | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/25 | 0/17
Other Adverse Events (participants affected / at risk) | 8/20 | 9/25 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acamprosate (N=20) | Naltrexone (N=25) | Placebo (N=17)
Fatigue (General disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0
Diaherrea (Gastrointestinal disorders) | 2 | 0 | 0
Decreased libido (Psychiatric disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No